CLINICAL TRIAL: NCT04616352
Title: Effect of Inappropriate Therapy With Cefuroxime in Adult Patients Hospitalized With Pyelonephritis
Brief Title: Cefuroxime Resistance in Pyelonephritis
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Jorge Alberto Cortes Luna, Primary investigator, Universidad Nacional de Colombia
Other Study IDs: ivucef001
Record Dates: First submitted 2020-10-18; First posted 2020-11-04 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Urinary Tract Infections
Keywords: pyelonephritis; urinary tract infections, complicated; cefuroxime; cephalosporins; Escherichia coli; Drug Resistance, Microbial
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis; Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Resistance to cefuroxime — Non susceptibility in vitro testing

SUMMARY:
Resistance to empirical antibiotic treatment has resulted in increased mortality and morbidity in serious infections caused by certain common resistant pathogens in the community. The risk for increased mortality has been also the motivation for recent guidelines that suggest early empirical antimicrobial treatment with broad spectrum antibiotics within a few hours of suspecting sepsis, regardless of the potential microorganism or infection focus. Resistance to second-generation cephalosporins among patients with community-acquired urinary tract infection by E. coli has exceeded 20% in an increasing number of institutions and communities, without being clear about the impact of such resistance on the effectiveness of treatment. This is especially important in urinary infections, since, in general, mortality is very low. We expect to establish if there is a relationship between inappropriate empirical therapy and morbidity (in terms of length of stay or readmission) among hospitalized patients with pyelonephritis treated with empirical cefuroxime therapy to help to define the need for a change in the current guidelines. These guidelines will have application not only in Colombia, but also in other countries in Latin America or other countries that still use this empirical therapy. It will also define the need for use of broader spectrum antibiotics in this clinical scenario.

DETAILED DESCRIPTION:
Objectives:

1. Establish the relationship between inappropriate empirical cefuroxime therapy in adult patients hospitalized with pyelonephritis and hospital stay.
2. Establish the relationship between inappropriate empirical cefuroxime therapy in adult patients hospitalized with pyelonephritis and readmission due to pyelonephritis.
3. Establish the relationship between inappropriate empirical therapy with cefuroxime in adult patients hospitalized with pyelonephritis and the time to readmission caused pyelonephritis.

The investigators proposed a retrospective cohort of hospitalized pyelonephritis patients with empirical antimicrobial management with cefuroxime in one institution of third complexity level. Exposure is understood as resistance to cefuroxime, that is, the impact of inappropriate empirical cefuroxime therapy on patients receiving this antibiotic. Patients who are admitted to the cohort had the diagnosis of pyelonephritis and were hospitalized for intravenous antimicrobial treatment and are followed up to the following outcomes: hospital discharge, or readmission due to pyelonephritis to the same or another institution of the insurance network.

The study will be conducted following the Good Clinical Practices for Research and approval by the Research Ethics Committee (REC) or Investigation Research Boards (IRB) of the participating institutions. The clinical information will be collected through online forms based on the information in the electronic medical record. Microbiological information will be taken from clinical laboratory reports (Whonet ver 5.5., WHO). The accuracy of the information collected will be verified by evaluating 100% of the formats. A pilot test will be carried out after approval by the IRB (25 february, 2020). The information will be stored anonymously, discarding from the database personal information of the patient that might allow the identification. Variables collected from the Electronic Medical Record include demographic, clinical (comorbidities, clinical status) and microbiological information. Other variables include time to change antibiotic (if done) and time of use of antibiotic. Information for the outcomes proposed include length of stay (in days), readmission (new admission because of pyelonephritis in the following 30 days after the first episode), and time to readmission (in days).

A propensity score matching will be performed to diminish the risk of selection bias and unbalanced subjects. Alternatively, and inverse probability treatment weighting can be used to balance the variables included. Both models will be constructed using a logistic regression for the probability of cefuroxime resistant. Final comparison between the exposed population and control population will be done using survival curves for the time to hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinical diagnosis of pyelonephritis.
* Antibiotic treatment with cefuroxime.
* Urine culture positive for Escherichia coli

Exclusion Criteria:

* Use of antibiotic for less than 24 hours.
* Not availability of antimicrobial susceptibility testing.
* Use of urinary catheter for more than 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiens with ≥ 18 years with a clinical diagnosis of community acquired pyelonephritis that require hospitalization and with positive culture for Escherichia coli.
Sampling Method: Non-Probability Sample
Enrollment: 973 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Time to hospital discharge | Up to 30 days
  Time since admission to hospital discharge
Readmission | Up to 30 days after discharge
  Proportion of patients admitted to hospital because of new episode of urinary tract infection
Time to readmission | Up to 30 days after discharge
  Time since discharge to readmission

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Cortes, MD, Principal Investigator — Univesidad Nacional de Colombia
Locations (1):
- Clínica Reina Sofía, Bogotá, DC, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nocua-Baez LC, Cortes JA, Leal AL, Arias GF, Ovalle-Guerro MV, Saavedra-Rojas SY, Buitrago G, Escobar-Perez JA, Castro-Cardozo B. [Antimicrobial susceptibility profile in urinary pathogens causing community-acquired infections in diabetic patients in Colombia]. Biomedica. 2017 Sep 1;37(3):353-360. doi: 10.7705/biomedica.v37i3.3348. Spanish. PMID 28968012
- [Background] Leal AL, Cortes JA, Arias G, Ovalle MV, Saavedra SY, Buitrago G, Escobar JA, Castro BE; GREBO. [Emergence of resistance to third generation cephalosporins by Enterobacteriaceae causing community-onset urinary tract infections in hospitals in Colombia]. Enferm Infecc Microbiol Clin. 2013 May;31(5):298-303. doi: 10.1016/j.eimc.2012.04.007. Epub 2012 Jun 15. Spanish. PMID 22703702